CLINICAL TRIAL: NCT02379533
Title: Effects of Home-based or Center-based Aerobic Exercise on Physical Function, Nutritional Status Ans Cardiopulmonary Parameters in Patients With Chronic Kidney Disease
Brief Title: Effects of Home-based or Center-based Aerobic Exercise in Patients With Chronic Kidney Disease
Acronym: HBCKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Lilian Cuppari, PhD, Affiliate Professor, Federal University of São Paulo
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009/14786-0
Record Dates: First submitted 2015-02-11; First posted 2015-03-05 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Renal Failure; Obese
MeSH Terms: conditions — Kidney Failure, Chronic; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sedentary control (No Intervention)
- Home-based aerobic exercise (Experimental): The training program will be conducted in accordance with the recommendations of the American College of Sports Medicine. All training sessions will be preceded by stretching of large muscle groups and heating (5 minutes) and at the end by cool down and stretching (5 minutes). The program will consist of 24 weeks with three sessions per week on alternate days. The aerobic training will be continuous, with an increment of 10 minutes in duration every 4 weeks. The intensity will be prescribed according to ventilatory threshold, characterized by the highest intensity of physical exertion fully maintained by aerobic energy pathways. The intensity control was done by means of the heart rate value obtained at ventilatory threshold. The home-based exercise group exercise at home with telephone follow-up weekly and once a month will be held at the training center under the supervision of a physical education teacher.
  Interventions: Other: Aerobic exercise
- Center-based aerobic exercise (Active Comparator): The training program will be conducted in accordance with the recommendations of the American College of Sports Medicine. All training sessions will be preceded by stretching of large muscle groups and heating (5 minutes) and at the end by cool down and stretching (5 minutes). The program will consist of 24 weeks with three sessions per week on alternate days. The aerobic training will be continuous, with an increment of 10 minutes in duration every 4 weeks. The intensity will be prescribed according to ventilatory threshold, characterized by the highest intensity of physical exertion fully maintained by aerobic energy pathways. The intensity control was done by means of the heart rate value obtained at ventilatory threshold. However, a group exercise held in the center on a treadmill with the direct supervision of a physical education teacher.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise
  Arms: Center-based aerobic exercise; Home-based aerobic exercise

SUMMARY:
Patients will be randomly assigned to perform the training program in center or home-based . The training program will be conducted in accordance with the recommendations of the American College of Sports Medicine. All training sessions will be preceded by stretching of large muscle groups and heating (5 minutes) and at the end by cool down and stretching (5 minutes). The program will consist of 24 weeks with three sessions per week on alternate days. The aerobic training will be continuous, with an increment of 10 minutes in duration every 4 weeks. The intensity will be prescribed according to ventilatory threshold, characterized by the highest intensity of physical exertion fully maintained by aerobic energy pathways. The intensity control was done by means of the heart rate value obtained at ventilatory threshold.

Both groups receive the same intervention. However, a group exercise held in the center on a treadmill with the direct supervision of a physical education teacher. The other group will exercise at home with telephone follow-up weekly and once a month will be held at the training center under the supervision of a physical education teacher.

It will also constituted a control group remain without performing any activity during the study period. After 24 weeks patients receive the same advice the team conducting the training at home.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals with chronic kidney disease stages 3 or 4 disease;
* Both genders;
* Age between 30 and 65 years;
* Overweight (BMI> 25 kg/m2);
* With a negative stress test.

Exclusion Criteria:

* Patients with chronic obstructive pulmonary disease,
* class IV heart failure,
* myocardial infarction within the last 6 months,
* decompensated hypertension (systolic blood pressure> 180 mmHg or diastolic> 110 mmHg in the last 6 months),
* uncontrolled cardiac arrhythmia,
* decompensated diabetes mellitus (glycated hemoglobin> 8.0%),
* unstable angina,
* infectious processes in the last 3 weeks;
* begin use of erythropoietin or with hemoglobin <11g/L.
* use of beta-blocker medication

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary capacity | 24 weeks
  The test began with a fixed inclination of 1%. The initial velocity was 2 km/h during the first three minutes with increments of 0.5km/h every minute until the patient reaches physical exhaustion. The ventilatory variables were measured using a gas analyzer. The highest oxygen uptake obtained during the last stage reached was considered the peak oxygen uptake. The ventilatory threshold was determined as the stage preceding the first occurrence of the exponential increase in ventilation, increase in the ventilatory equivalent for oxygen and increase in expired fraction of oxygen. The respiratory compensation point was determined as the stage preceding the second occurrence of the exponential increase in ventilation, increase in the ventilatory equivalent for carbon dioxide and decrease in end-tidal carbon dioxide. Data were analyzed by the average of 20 seconds.
Functional capacity (walk, sit-stand, arm curl, sit-reach, back scratch, timed up and go) | 24 weeks
  Functional capacity was assessed using a variety of objective measures. These included six-minute walk test (maximal distance walked along an internal corridor during six minutes), two-minute step test (maximal number of steps achieved in stationary walking during two minutes, used to quantifying the aerobic power), sit-to-stand test (maximal sit to stand cycles achieved in 30 seconds, used to quantifying the muscular endurance of the legs), arm curl test (maximal number of arm curl cycles in 30 seconds, used to quantifying the muscular endurance of the arms), sit and reach test (maximal distance achieved in the Wells bench, used to quantifying the general flexibility), back scratch test (maximum amplitude of the arms used to quantifying the arms flexibility) and time up and go test (shorter time to rise from a chair, walk three meters and sit back, used to quantifying the functional mobility).

SECONDARY OUTCOMES:
Quality of life | 24 weeks
  The Short-Form Health Survey (SF-36) questionnaire was applied to assess the quality of life. The scores for each domain range from 0 to 100%. The higher scores define a better quality of life. The questionnaire was applied individually in a clear and quiet room with the patient rested.
sleep quality (PSQI) | 24 weeks
  The PSQI assesses the quality of sleep for the last month of the interview. The questionnaire has 19 questions that comprise seven assessment components: quality of sleep, latency, duration, efficiency, nocturnal sleep disturbances, use of sleep medication and daytime sleepiness. Each component receives a score from 0 to 3, in a way that the final score can range between 0 and 21. The higher the score, the worse the quality of sleep, and scores higher than five indicate sleep disturbances.
blood pressure | 24 weeks
  Blood pressure and resting heart rate were measured before the cardiopulmonary exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Cuppari, PhD, Principal Investigator — Federal University of São Paulo; Danilo T Aoike, MSc, Principal Investigator — Federal University of São Paulo

REFERENCES:
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Gomes TS, Aoike DT, Baria F, Graciolli FG, Moyses RMA, Cuppari L. Effect of Aerobic Exercise on Markers of Bone Metabolism of Overweight and Obese Patients With Chronic Kidney Disease. J Ren Nutr. 2017 Sep;27(5):364-371. doi: 10.1053/j.jrn.2017.04.009. Epub 2017 Jun 9. PMID 28606422